CLINICAL TRIAL: NCT01364714
Title: Biomechanical Properties in ICU Survivors 12-month After Discharge
Brief Title: Biomechanical Properties in Intensive Care Unit (ICU) Survivors 12-month After Discharge
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jesper Poulsen, MD, Rigshospitalet, Denmark
Other Study IDs: 2008-120-25298
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Intensive Care (ICU) Myopathy
Keywords: ICU acquired weakness
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- ICU survivors: Male ICU survivors 12 month after discharge
- Controls: Age and gender matched controls

SUMMARY:
Intensive care unit (ICU) admission is associated with muscle weakness and ICU survivors report persevering limitation of physical capacity for years after discharge. Limited information is available about the underlying biomechanical properties responsible for this muscle function impairment.

ELIGIBILITY:
Inclusion Criteria:

* ICU length of stay > 72 hours
* Informed consent

Exclusion Criteria:

* BMI>30
* Neuromuscular or psychiatric disease

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ICU survivors 12 months after discharge compared to age and gender matched controls
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Biomechanics and Motor Control Laboratory, Department of Exercise and Sport Sciences, University of Copenhagen, Copenhagen, Denmark